CLINICAL TRIAL: NCT02106702
Title: Navigator-Enhanced Case Management for HIV-Infected Jail Inmates Reentering the Community
Brief Title: The Navigator Project
Acronym: NAV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: San Francisco Jail Health Services - HIV and Integrated Services (Unknown); San Francisco Pretrial Diversion Project (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R01DA027209 (NIH)
Record Dates: First submitted 2014-04-01; First posted 2014-04-08 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: HIV
Keywords: HIV; detention; substance abuse
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- FAP counseling (Active Comparator): Control arm utilizing the standard of care: access to services provided by the Forensic AIDS Project for up to 90 days after release
  Interventions: Behavioral: Forensic AIDS Project
- Navigator enhanced case-management (Experimental): Experimental arm: access to Navigator enhanced case-management services for one year after release
  Interventions: Behavioral: Navigator enhanced case-management

INTERVENTIONS:
Behavioral: Navigator enhanced case-management — Patient navigators are non-clinical, paraprofessional peers who are HIV-infected and have lifetime histories of detention and substance abuse. Working with the patient, they facilitate adherence to a comprehensive care plan designed to address clients' multiple risks and needs. Patients have access to Navigator services for one year after study enrollment.
  Arms: Navigator enhanced case-management
Behavioral: Forensic AIDS Project — The Forensics AIDS Project provides primary care to HIV-infected detainees, as well as up to 90 post-release case-management services which include discharge planning.
  Arms: FAP counseling

SUMMARY:
Each year, there are over 600 unduplicated HIV-infected persons incarcerated in the San Francisco jail. Two thirds of those released with HIV-focused discharge planning are reincarcerated within one year. More than half of HIV-infected jail inmates are diagnosed with mental health conditions severe enough to require medication and a similar proportion report substance use disorders at the time of detention. While some community-based services exist, there remains a critical need to improve linkages to care and adherence to care plans for HIV-infected adults as they move between community and jail. The Navigator Project is a five-year randomized study that will test the effectiveness of an intensive enhanced case management intervention to reduce sex and drug-related HIV transmission risk; increase HIV medication adherence; reduce drug dependence; and reduce reincarceration.

ELIGIBILITY:
Inclusion Criteria:

* Detention in the San Francisco jail system
* Confirmed HIV infection
* Lifetime history of ever having met standardized criteria for drug or alcohol addiction
* Likely release back into San Francisco without transfer to another facility
* Agreement to work with Forensic AIDS Project to plan post-release care
* Able and willing to provide informed consent
* Not scheduled for release within 36 hours

Exclusion Criteria:

* Undocumented HIV status
* Inability to speak English or Spanish
* Unable or unwilling to provide informed consent
* Not under routine level of jail security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 271 (Actual)
Dates: Start 2010-02; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
substance use | 2 months, 6 months, 12 months
  change from baseline in self-reported drug and alcohol use, measured by a survey tool, and actual use of five drugs (methamphetamine, cocaine, tetrahydrocannabinol, opiates, and benzodiazepines), measured by a urine screen, at three time points each
recidivism | 12 months
  number of times re-detained during the twelve-month study period, collected from jail records

SECONDARY OUTCOMES:
sexual risk behavior | 2 months, 6 months, 12 months
  change from baseline in self-reported sexual risk behaviors, measured by a survey tool at three time points after the initial detention
adherence to HIV medications | 2 months, 6 months, 12 months
  change from baseline in self-reported adherence (as a %) to antiretroviral therapy, measured by a survey tool at three time points after the initial detention

OTHER OUTCOMES:
housing | 2 months, 6 months, 12 months
  change from baseline in self-reported housing status, measured by a survey tool at three time points after the initial detention
medical coverage | 2 months, 6 months,12 months
  change from baseline in self-reported insurance coverage, measured by a survey tool at three time points after the initial detention, and use of community health services and jail health services, measured continuously via a community database for 12 months after the initial detention
needle use | 2 months, 6 months, 12 months
  change from baseline in self-reported needle-use and needle-sharing, measured by a survey tool at three time points after the initial detention

CONTACTS AND LOCATIONS:
Overall Officials: Janet J Myers, PhD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- Tenderloin Clinical Research Foundation, San Francisco, California, United States